CLINICAL TRIAL: NCT00657475
Title: A Prospective Study of Coronary Artery Bypass Graft and/or Aortic Valve Replacement With Conventional Versus Half Heparin Dose Under Closed and Coated Extra Corporeal Circulation System (MECC) - APPACHES Study.
Brief Title: Coronary Bypass and Artotic Leaflet Surgery : Heparin Low Dose vs Full Dose
Acronym: APPACHES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUBX 2007/19
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Cardiac Surgery; Extracorporeal Circulation
Keywords: Heparin low dose; Inflammation; Blood loss
MeSH Terms: conditions — Inflammation; Hemorrhage | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Cardiac surgery with Mini Extra Corporeal Circulation (MECC). Heparin low dose (150 UI/Kg).
  Interventions: Drug: Heparin Low Dose
- 1 (Active Comparator): Cardiac surgery with Mini Extra Corporeal Circulation (MECC). Heparin Full Dose (300 UI/Kg)
  Interventions: Drug: Heparin Full Dose

INTERVENTIONS:
Drug: Heparin Low Dose — Loading heparin dose of 150 IU / kg to achieve an ACT (activating clotting time) target more than 240 seconds.
  Arms: 2
Drug: Heparin Full Dose — Loading heparin dose of 300 IU / kg to achieve an ACT (activating clotting time) target more than 400 seconds.
  Arms: 1

SUMMARY:
The purpose of this study is to demonstrate superiority on postoperative bleeding from the use of a heparin half dose compared to a conventional dose, under mini-extra corporeal circulation, without increased risk to the patient.

DETAILED DESCRIPTION:
Usually management of conventional extra corporeal circulation takes place under a loading heparin dose of 300 IU / kg to achieve an ACT (activating clotting time) target more than 400 seconds. This empirical approach based on patient weight date from the 1960's and does not take into account materials improvement and different individual sensitivities; several studies have demonstrated than a result at least as effective could be obtained with heparin lower doses, and without increasing thromboembolic morbid events for patients.

Patients are randomly assigned into one of 2 groups one day before surgery. First group receive unfractionated heparin conventional dose during the MECC, second group receive half of the conventional dose. All surgery is performed by the same team and using same equipment. Regular blood tests are carried out before, during and after surgery. Blood loss, transfusion needs, rhythm disorders, stay duration in intensive care and total hospitalization length is finally reported. The follow-up period through the 30th postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* single or multiple coronary bypass
* written and informed consent
* repair or replacement of artic leaflet
* platelet suppressive agents stopped since at least 7 days
* anticoagulants stopped since at least 3 days

Exclusion Criteria:

* Thoracic surgery antecedent
* ASA 4
* carotid stenosis > 75%
* Hb < 10,5 g/l
* chronic hepatic failure
* thromboembolic antecedent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2008-06; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Blood loss | Peroperative and postoperative until redon's suction drainage ablation

SECONDARY OUTCOMES:
Blood transfusion | Per & postoperative
Use of intropic drugs (posology) | Postoperative
Kidney function(urea, creatininemia) | Postoperative
Peroperative hemodynamic data | Peroperative

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ROQUES, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Cardiac Surgery Dpt (University Hospital), Bordeaux, France